CLINICAL TRIAL: NCT01329471
Title: Functional Role of RUNX1 Mutations in the Etiology of Acute Myeloid Leukemia (AML)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Dr. Ofer Fainaru, Hillel Yaffe Medical Center
Other Study IDs: HYMC-16-2011
Record Dates: First submitted 2011-03-10; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Umbilical cord blood

SUMMARY:
The purpose of this study is to elucidate the role of RUNX1 in Acute Myeloid Leukemia (AML), in particular, the transcriptional regulation of genes by mutated forms of this protein. This research will study the effect of mutations found in AML patients

DETAILED DESCRIPTION:
The RUNX1 gene, located at chromosomal band 21q22, is a transcription factor, crucial for hematopoiesis and the generation of hematopoietic stem cells in the embryo. RUNX1 is the most frequent target for chromosomal translocation in leukemia. In addition, point mutations in the RUNX1 gene have been found to constitute an important mode of genetic alteration in development of leukemia. Recent publications stressing the clinical need for implementing RUNX1 point mutations as both a diagnostic and unfavorable prognostic marker of AML, have aroused particular interest in the functional role of RUNX1 in this disease.

In order to pinpoint specific RUNX1 target genes involved in pre-leukemic transformation or exacerbation of existing leukemia, the investigators plan to compare expression profiles from human hematopoietic progenitors overexpressing a mutated form of RUNX1with controls (RUNX1 wild-type and knocked-down). In this study the investigators intend to collect blood, after receiving informed consent, from umbilical cords of neonates born vaginally, in order to isolate CD34+ hematopoietic progenitors. Human umbilical cord blood contains relatively high numbers of CD34+ cells, which may be frozen directly after collection and used as a source of progenitor cells for further culture or direct analysis.

ELIGIBILITY:
Inclusion Criteria:

* Consenting women who have had full-term birth

Exclusion Criteria:

* Systemic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female hospital patients
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Performance of expression arrays on transfected CD34+ cells | One year
  Performance of expression arrays on transfected CD34+ cells (derived from human cord blood), expecting differential gene expression between the wild type RUNX1-transfected cells and mutated RUNX1-transfected cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel